CLINICAL TRIAL: NCT04496531
Title: Examining the Efficacy of Non-invasive Neuromodulation in Reducing Symptoms of Multiple Sclerosis - a Pilot Study
Brief Title: Efficacy of PoNS in Reducing Symptoms of Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helius Medical Inc (Industry)
Collaborators: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS Pilot - Leonard, et al
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Fourteen MS patients, seven each in an active and a sham stimulation group, participated.
  Participants received intensive physical therapy and working memory training for 14 weeks. Functional magnetic resonance imaging (fMRI) using motor imagery and working-memory tasks were completed prior to and following therapy, as were sensory organization tests (SOT), motor performance measures, and neuropsychological assessment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Therapists and other personnel (MR technicians, SOT and DGI administrators, Neuropsychologists etc.) were not informed as to which group a subject belonged. In order to maintain this blinding, both subjects and therapists were instructed not to discuss any details of the stimulus sensation with each other. Additionally, all subjects were instructed not to adjust the stimulus intensity in the presence of therapists. All questions about device use or the stimulation were to be addressed only to the PI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Active group members use a device providing perceivable electrical stimulation
  Interventions: Device: Portable Neuromodulation Stimulator
- Sham (Sham Comparator): Group members use a device providing a non-perceivable stimulus
  Interventions: Device: Portable Neuromodulation Stimulator

INTERVENTIONS:
Device: Portable Neuromodulation Stimulator
  Other Names: PoNS

SUMMARY:
The purpose of this pilot study is to determine whether a program involving both in-lab and at-home training using cranial nerve stimulation (CN-NINM) delivered via the tongue can reduce symptoms of multiple sclerosis (MS) and improve movement control and therefore provide ground work for a controlled clinical trial. The effects of the stimulation will be measured using a variety of standardized tests of movement control and cognitive function, functional brain imaging, and MS-specific surveys of your quality of life.

DETAILED DESCRIPTION:
Fourteen MS patients, seven each in an active and a sham stimulation group are expected to participate.

Participants will receive intensive physical therapy and working memory training for 14 weeks.

Functional magnetic resonance imaging (fMRI) using motor imagery and working-memory tasks will be completed prior to and following therapy, as will be sensory organization tests (SOT), motor performance measures, and neuropsychological assessment.

Prior to the start of CN-NINM training, each participant will undergo baseline evaluations including structural and fMRI, balance tests (SOT), Dynamic Gait Index (DGI), neuropsychological assessment (Handedness; Wechsler Abbreviated Scale of Intelligence (WASI) Vocabulary and Matrix Reasoning; California Verbal Learning Test (CVLT)-11; D-Kefs Trails, Color/Word and Verbal Fluency; Tower of London Second Edition; Ruff 2 and 7; Wechsler Adult Intelligence Scale Fourth Edition (WAIS-IV) Letter-Number sequencing, Coding and Symbol Search; Paced Auditory Serial Addition Test (PASAT); Leonard Tapping; and Grooved Pegboard). In addition, the MS Impairment Scale, Fatigue Impact Scale, Cognitive Function Inventory for MS, and Beck Depression and Anxiety questionnaires will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing/remitting or secondary progressive MS with balance and gait problems;
* Recent EDSS score of 3.0 - 6.0;
* Provided informed consent and willing to participate

Exclusion Criteria:

* Use of tobacco products;
* Oral health problems including abrasions, cuts, cold sores, piercings, or tissue inflammation in the oral cavity;
* Baseline EDSS >6.

Ages: 28 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index | 14 weeks
  Scores are based on a 4-point scale where: 3 = No gait dysfunction; 2 = Minimal impairment; 1 = Moderate impairment; and 0 = Severe impairment. The highest possible score was 24 points. Tasks include: Steady state walking; Walking with changing speeds; Walking with head turns both horizontally and vertically; Walking while stepping over and around obstacles; Pivoting while walking; and Stair climbing.

IPD SHARING:
Plan to Share IPD: No